CLINICAL TRIAL: NCT02777034
Title: Short-Term Outcomes of Laparoscopy Combined With Enhanced Recovery Pathway After Ileocolon Resection for Crohn's Disease
Brief Title: Laparoscopy Combined With Enhanced Recovery Pathway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhou, Doctor, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SRRSH20160427-001
Record Dates: First submitted 2016-05-13; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Crohn's Disease
Keywords: Laparoscopy; Enhanced Recovery; Fast-track
MeSH Terms: conditions — Crohn Disease | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Recovery (Experimental): Preoperative protocols：Multidisciplinary patient information、no bowel preparation、no fasting（drink 10% glucose 1000 at 21：30 night before the surgery）.
  Intraoperative protocols：Laparoscopic standardized technique、fluid restriction (max 500 ml/h)、no abdominal drains.
  Postoperative protocols：no nasogastric tube、early solid dietary intake and mobilization、urinary catheter removal on postoperative day 1、restrictive fluid management（<2000ml/d）.
  Interventions: Other: ER
- Unenhanced Recovery (Other): Preoperative protocols：Patient information、Mechanical bowel preparation、Fasting since midnight before operation.
  Intraoperative protocols：Laparoscopic standardized technique、fluid overload (over 500 ml/h) 、place abdominal drains.
  Postoperative protocols：no nasogastric tube、mobilization from postoperative day 1、fluids and solids intake after first passage of stool、Urinary catheter removal on postoperative day 2/3、no restrictive fluid management（>2000ml/d）.
  Interventions: Other: UR

INTERVENTIONS:
Other: ER — Preoperative protocols：Multidisciplinary patient information、no bowel preparation、no fasting（drink 10% glucose 1000 at 21：30 night before the surgery）.
  Intraoperative protocols：Laparoscopic standardized technique、fluid restriction (max 500 ml/h)、no abdominal drains.
  Postoperative protocols：no nasogastric tube、early solid dietary intake and mobilization、urinary catheter removal on postoperative day 1、restrictive fluid management（<2000ml/d）.
  Other Names: Enhanced Recovery
  Arms: Enhanced Recovery
Other: UR — Preoperative protocols：Patient information、Mechanical bowel preparation、Fasting since midnight before operation.
  Intraoperative protocols：Laparoscopic standardized technique、fluid overload (over 500 ml/h) 、place abdominal drains.
  Postoperative protocols：no nasogastric tube、mobilization from postoperative day 1、fluids and solids intake after first passage of stool、Urinary catheter removal on postoperative day 2/3、no restrictive fluid management（>2000ml/d）.
  Other Names: Un-Enhanced Recovery
  Arms: Unenhanced Recovery

SUMMARY:
Laparoscopy combined with an enhanced recovery pathway versus laparoscopy combined with a traditional recovery pathway after ileocolon resection for Crohn's Disease.

DETAILED DESCRIPTION:
Thirty patients with CD of ileocolon will be randomly assigned to two groups.One group is ERP group which include no bowel preparation nor fasting, no abdominal drains, early removal of urinary catheter, early solid dietary intake and mobilization and restrictive fluid management.In the end,we can compare the time to first flatus、time to first flatus 、postoperative length of stay postoperative hospital expense、complication grade readmission within 30 days of discharge between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years≤aged≤75 years) were included if they had histologically or radiographic proven CD with disease localized to the terminal ileum with or without ascending colon involvement.

Exclusion Criteria:

* Those patients were excluded：previous bowel resection or strictureplasty, preoperative radiological evidence of large phlegmons/abscesses/enteric fistulas (assessed by magnetic resonance imaging or computed tomography), emergency surgery, and anesthesiological contraindications to laparoscopy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The time of Flatus and Defecation | 0-10 days

SECONDARY OUTCOMES:
The time of liquid diet and semiliquid diet | 0-10 days

OTHER OUTCOMES:
Postoperative complications | 0-10 days
Postoperative hospitalization cost | 0-10 days
Hospital readmission rates | 0-30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhou, Doctor, Study Chair — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Spinelli A, Bazzi P, Sacchi M, Danese S, Fiorino G, Malesci A, Gentilini L, Poggioli G, Montorsi M. Short-term outcomes of laparoscopy combined with enhanced recovery pathway after ileocecal resection for Crohn's disease: a case-matched analysis. J Gastrointest Surg. 2013 Jan;17(1):126-32; discussion p.132. doi: 10.1007/s11605-012-2012-5. Epub 2012 Sep 5. PMID 22948838
- [Result] Andersen J, Kehlet H. Fast track open ileo-colic resections for Crohn's disease. Colorectal Dis. 2005 Jul;7(4):394-7. doi: 10.1111/j.1463-1318.2005.00788.x. PMID 15932565
- [Result] Veenhof AA, Vlug MS, van der Pas MH, Sietses C, van der Peet DL, de Lange-de Klerk ES, Bonjer HJ, Bemelman WA, Cuesta MA. Surgical stress response and postoperative immune function after laparoscopy or open surgery with fast track or standard perioperative care: a randomized trial. Ann Surg. 2012 Feb;255(2):216-21. doi: 10.1097/SLA.0b013e31824336e2. PMID 22241289
- [Derived] Zhu Y, Xiang J, Liu W, Cao Q, Zhou W. Laparoscopy Combined with Enhanced Recovery Pathway in Ileocecal Resection for Crohn's Disease: A Randomized Study. Gastroenterol Res Pract. 2018 Nov 11;2018:9648674. doi: 10.1155/2018/9648674. eCollection 2018. PMID 30534152